CLINICAL TRIAL: NCT02286050
Title: Auswirkung Eines CF Nursing-Programms Auf Das Krankheitsmanagement Und Die Erfahrungen Der Behandlung Von Patientinnen Und Patienten
Brief Title: Effect of a Nursing Program for Patients With Cystic Fibrosis on Disease Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SNCTP000000179
Record Dates: First submitted 2014-10-27; First posted 2014-11-07 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

ARMS (1):
- CF Nursing Intervention (Experimental)
  Interventions: Other: CF Nursing Program

INTERVENTIONS:
Other: CF Nursing Program

SUMMARY:
The purpose of this study is to evaluate the effect of a nursing program in patients with cystic fibrosis.

DETAILED DESCRIPTION:
All patients living with cystic fibrosis will be asked by questionnaire before (November 2014) and after (September 2016) the implementation of the program about their satisfaction with treatment, trust in the CF-Team, adherence, self-efficacy, treatment burden and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Cystic Fibrosis

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-11; Primary Completion 2017-02 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Difference between baseline patient satisfaction and month 22 | month 22
  Self-reported patient satisfaction will be measured with a newly developped questionnaire.

SECONDARY OUTCOMES:
Difference between baseline adherence and month 22 | month 22
  Self-reported adherence to therapy will be measured with the Medication Adherence Report Scale (MARS) and a newly developped questionnaire.
Difference between baseline self-efficacy and month 22 | month 22
  Self-reported self-efficacy to master the the therapeutic regimen will be measured with a newly developped questionnaire.
Difference between baseline treatment burden and month 22 | month 22
  Self-reported treatment burden will be measured wiht a subscale of the CFQ-R.
Difference between baseline trust and month 22 | month 22
  Self-reported trust will be measured with the short version of the Wake Forest Trust Scale.
Difference between baseline information need and month 22 | month 22
  Information needs will be assessed with a subscale of the PICKER-questionnaire for patients with CF.

OTHER OUTCOMES:
Difference between baseline QoL and month 22 | month 22
  Self-reported QoL will be measured with the Cystic Fibrosis Questionnaire - revised (CFQ-R) and the VAS of the European Quality of Life Instrument - 5 dimensions (EQ-5D VAS).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Switzerland